CLINICAL TRIAL: NCT01023061
Title: Phase II Trial of Radiation With Androgen Deprivation: Abiraterone Acetate, Prednisone and Luteinizing Hormone Releasing Hormone Agonist Prior to Radiation Therapy
Brief Title: Abiraterone Prednisone and Hormonal Therapy Before and During Radiation Therapy in Localized Prostate Cancer
Acronym: RAD1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bruce Montgomery, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7048; NCI-2009-01346 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 7048 - AbiRAD; 7048 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Adenocarcinoma of the Prostate; Stage II Prostate Cancer; Stage III Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone; Leuprolide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (antihormone therapy and radiation therapy) (Experimental): Patients receive abiraterone acetate and prednisone daily for 24 weeks. Patients also receive leuprolide acetate or goserelin in weeks 1 and 13. Patients undergo external beam radiotherapy starting in week 15 for 8.5 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: abiraterone acetate; Drug: prednisone; Drug: leuprolide acetate; Other: laboratory biomarker analysis; Radiation: external beam radiation therapy; Drug: goserelin acetate

INTERVENTIONS:
Drug: abiraterone acetate — Given PO
  Other Names: Zytiga
Drug: prednisone — Given PO
  Other Names: DeCortin; Deltra
Drug: leuprolide acetate — Given via injection
  Other Names: Enantone; Lupron; Lupron Depot
Other: laboratory biomarker analysis — Correlative study
Radiation: external beam radiation therapy — Undergo radiotherapy
Drug: goserelin acetate — Given via injection
  Other Names: Zoladex

SUMMARY:
This phase II trial studies the side effects and how well abiraterone acetate, prednisone, and leuprolide acetate or goserelin before and during radiation therapy works in treating patients with localized or locally advanced prostate cancer. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as abiraterone acetate, leuprolide acetate, and goserelin, may lessen the amount of androgens made by the body. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving abiraterone acetate and leuprolide acetate or goserelin before or together with radiation therapy may be an effective treatment for prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of abiraterone (abiraterone acetate) and prednisone with luteinizing hormone-releasing hormone agonist given as neoadjuvant and concurrent therapy with external beam radiation in patients with localized prostate cancer.

II. To determine whether pharmacologic suppression of the prostatic androgen axis by inhibition of androgen production with abiraterone can decrease tissue androgen levels to below those observed with gonadotropin-releasing hormone (GnRH) agonist suppression of testicular androgens.

SECONDARY OBJECTIVES:

I. To determine whether treatment with abiraterone acetate with luteinizing releasing hormone agonist will be more effective than agonist with bicalutamide in inducing inhibition of androgen-regulated gene expression and increased apoptotic cell death as assessed by immunohistochemistry, complementary deoxyribonucleic acid (cDNA) microarray analysis and reverse transcription-polymerase chain reaction (RT-PCR).

II. To evaluate time to prostate-specific antigen progression in patients treated with GnRH agonist with abiraterone acetate.

OUTLINE:

Patients receive abiraterone acetate orally and prednisone once daily for 24 weeks. Patients also receive leuprolide acetate or goserelin in weeks 1 and 13. Patients undergo external beam radiotherapy starting in week 15 for 8.5 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Patients must allow biopsy prior to neoadjuvant therapy and at the time of fiducial placement
* Written Authorization for Use and Release of Health and Research Study Information has been obtained
* Histologically proven adenocarcinoma of the prostate
* Patients must be candidates for short or long term androgen deprivation in combination with external beam radiotherapy (RT) based on the following criteria:

  * Intermediate Risk Disease: T2b/c, or Gleason 7, or Prostate Specific Antigen 10-20
  * High Risk Disease: Gleason 8-10, or Prostate specific antigen> 20, or T3/4
* Patients may not have received any prior pharmacologic therapy or radiation therapy (RT) for prostate cancer
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Karnofsky >= 60%
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the androgen axis will be determined following review of their case by the Principal Investigator
* White blood cell count: >= 3,000/mm^3
* Absolute granulocyte count: >= 1,000/mm^3
* Platelets: >= 100,000/mm^3
* Hemoglobin >= 10g/dL
* Potassium >= 3.5 mmol/L
* Serum creatinine: =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) < 2.5 x ULN
* Alanine transaminase (ALT) < 2.5 x ULN
* Total bilirubin: =< 1.5 x ULN (except for patients with documented Gilbert's disease)

Exclusion Criteria:

* Patients may not be receiving any investigational agents
* Concurrent enrollment in another clinical investigational drug or device study is prohibited
* The concurrent administration of other anticancer therapy, including cytotoxic or hormonal agents (except Luteinizing hormone releasing hormone agonists), or immunotherapy, is prohibited during neoadjuvant concurrent and adjuvant therapy
* Patients who are currently receiving active therapy for other neoplastic disorders will not be eligible
* Patients with histologic evidence of small cell carcinoma of the prostate will not be eligible
* Patients with hypogonadism or severe androgen deficiency as defined by serum testosterone less than 100 ng/dL will not be eligible
* History of pituitary or adrenal dysfunction
* Patients who are receiving any androgens, estrogens or progestational agents, or who received any of these agents within the 6 months prior to evaluation will not be eligible
* Patients who are taking drugs which affect androgen metabolism (e.g. spironolactone, ketoconazole, finasteride, dutasteride) will not be eligible
* Concomitant therapy with any of the following listed is prohibited: 5 alpha-reductase inhibitor (finasteride, dutasteride); ketoconazole, diethylstilbestrol, and other preparations such as saw palmetto thought to have endocrine effects on prostate cancer; radiopharmaceuticals such as strontium (89Sr) or samarium (153Sm); Aldactone, Spironol (spironolactone); estrogens, testosterone, progesterones, herbal medications
* Patients who received any of these agents within the 6 months prior to evaluation will be reviewed for eligibility by the Principal Investigator on a case by case basis
* Use of other investigational drug therapy for any reason is prohibited
* Patients with inflammatory bowel disease or other autoimmune conditions which might affect the radiated colon or rectum
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, cardiac arrhythmia which is symptomatic or requires active therapy, recent deep venous thrombosis, pulmonary emboli, cerebrovascular accident or ischemia will not be eligible
* Patients who have chronic active hepatitis or acute hepatitis will not be eligible
* Patients with dementia/psychiatric illness/social situations that would limit compliance with study requirements or would prohibit the understanding and/or giving of informed consent will not be eligible
* Patients with medical conditions, which, in the opinion of the investigators, would jeopardize either the patient or the integrity of the data obtained will not be eligible
* Uncontrolled hypertension within the screening period (systolic blood pressure [BP] >= 160 mmHg or diastolic BP >= 95 mmHg)
* Patients with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive therapy
* History of congestive heart failure of any severity
* Other active malignancy, except non-melanoma skin cancer and superficial bladder cancer
* History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study drug
* Patients with diabetes not controlled with diet alone (i.e. requiring insulin or oral hypoglycemics)
* Patients unwilling to use contraceptives while on study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Montgomery, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - MultiCare Regional Cancer Center - Tacoma, Tacoma, Washington

REFERENCES:
- [Background] Cho E, Mostaghel EA, Russell KJ, Liao JJ, Konodi MA, Kurland BF, Marck BT, Matsumoto AM, Dalkin BL, Montgomery RB. External beam radiation therapy and abiraterone in men with localized prostate cancer: safety and effect on tissue androgens. Int J Radiat Oncol Biol Phys. 2015 Jun 1;92(2):236-43. doi: 10.1016/j.ijrobp.2015.01.020. Epub 2015 Mar 12. PMID 25772183

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Antihormone Therapy and Radiation Therapy): Patients receive abiraterone acetate and prednisone daily for 24 weeks. Patients also receive leuprolide acetate or goserelin in weeks 1 and 13. Patients undergo external beam radiotherapy starting in week 15 for 8.5 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  abiraterone acetate: Given orally
  prednisone: Given orally
  leuprolide acetate: Given via injection
  laboratory biomarker analysis: Correlative study
  external beam radiation therapy: Undergo radiotherapy
  goserelin acetate: Given via injection
Period: Overall Study
Arm/Group | Treatment (Antihormone Therapy and Radiation Therapy)
Started | 24
Completed (2 patients enrolled but withdrew from study prior to receiving study therapy) | 22
Not Completed | 2
Not completed — Withdrawal prior to treatment | 2

BASELINE CHARACTERISTICS:
Population: Men with intermediate or high risk localized prostate cancer
Groups:
- Treatment (Antihormone Therapy and Radiation Therapy): Patients receive abiraterone acetate and prednisone for 24 weeks. Patients also receive leuprolide acetate or goserelin in weeks 1 and 13. Patients undergo external beam radiotherapy starting in week 15 for 8.5 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  abiraterone acetate: Given orally
  prednisone: Given orally
  leuprolide acetate: Given via injection
  laboratory biomarker analysis: Correlative study
  external beam radiation therapy: Undergo radiotherapy
  goserelin acetate: Given via injection
Arm/Group | Treatment (Antihormone Therapy and Radiation Therapy)
Number analyzed (Participants) | 24
Age, Continuous [Median (Standard Deviation); unit: years] | 61 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Acute and Chronic Grade 3 or Greater Toxicity as Evaluated Using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 3.0
Description: Incidence of acute and chronic grade 3 or greater toxicity as evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.0he distribution of time to late adverse events (observed severities of adverse events over time) will be estimated using the Kaplan-Meier method.
Time Frame: Up to 24 months after initiation of radiation therapy
Population: Treated patients
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Antihormone Therapy and Radiation Therapy): Patients receive abiraterone acetate PO and prednisone PO for 24 weeks. Patients also receive leuprolide acetate or goserelin in weeks 1 and 13. Patients undergo external beam radiotherapy starting in week 15 for 8.5 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  abiraterone acetate: Given PO
  prednisone: Given PO
  leuprolide acetate: Given via injection
  laboratory biomarker analysis: Correlative study
  external beam radiation therapy: Undergo radiotherapy
  goserelin acetate: Given via injection
Arm/Group | Treatment (Antihormone Therapy and Radiation Therapy)
Number analyzed (Participants) | 22
Participants | 6
Statistical Analysis 1: Comparison: Treatment (Antihormone Therapy and Radiation Therapy); Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.74

2. Primary Outcome: Levels of Dihydrotestosterone (DHT) and Testosterone in Prostate Biopsy Sample Assessed by Mass Spectrometry
Description: The levels from patients treated in this study will be compared to a control set of biopsies acquired from a separate but similar population of men with intermediate and high risk prostate cancer treated with three months of combined Luteinizing hormone releasing hormone agonist and bicalutamide as part of standard of care.
Time Frame: Week 12
Population: Treated patients with measurable tissue DHT
Measure: Median (90% Confidence Interval); unit: pg/mg
Arm/Group | Treatment (Antihormone Therapy and Radiation Therapy)
Number analyzed (Participants) | 22
pg/mg | 0.050 [0.050 to 0.050]

3. Secondary Outcome: Median Time to Prostate Specific Antigen Progression
Description: Defined as the date of an increase of 2ng/mL or more above the Prostate specific antigen nadir achieved after completion of radiation with the date of progression defined as the date on which that value was measured. Distribution of time-to-event variables will be estimated using the Kaplan-Meier product-limit method. Estimated with two-sided 95% confidence intervals.
Time Frame: 6 months
Population: Treated patients
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Treatment (Antihormone Therapy and Radiation Therapy)
Number analyzed (Participants) | 22
years | 5 (1)

ADVERSE EVENTS:
Time Frame: Median follow-up 21 months
Description: Tracked grade 1 and 2 toxicities >10% and grade 3 toxicities that were either possibly or probably related to radiation, abiraterone or prednisone, or Luteinizing hormone releasing hormone agonist.
Arm/Group | Treatment (Antihormone Therapy and Radiation Therapy)
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 19/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Antihormone Therapy and Radiation Therapy) (N=22)
Lymphopenia (Blood and lymphatic system disorders) | 19 (19)
Hypertension (Cardiac disorders) | 8 (8)
ALT and AST: increased (Metabolism and nutrition disorders) | 7 (7)
fatigue (General disorders) | 15 (15)
hypokalemia syndrome (Investigations) | 12 (12)
Hot flashes (Vascular disorders) | 15 (15)
Hyperbilirubinemia (Hepatobiliary disorders) | 5 (5)
insomnia (General disorders) | 3 (3)
erectile dysfunction (Reproductive system and breast disorders) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 9 (9)
urinary tract discomfort (Renal and urinary disorders) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No